CLINICAL TRIAL: NCT00387335
Title: Phase II Study of Sunitinib Malate in Head and Neck Squamous Cell Carcinoma
Brief Title: Sunitinib in Treating Patients With Recurrent and/or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00214; NCI-2009-00214 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000504024; 7738 (Other: University of Chicago); 7738 (Other: CTEP); N01CM62201 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2012-12

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Sunitinib

ARMS (1):
- Arm I (Experimental): Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with recurrent and/or metastatic head and neck cancer. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the overall response rate of patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck treated with sunitinib malate.

II. Determine the toxicity of this drug in these patients. III. Determine the feasibility of administering this drug to patients with ECOG performance status 2 (cohort B).

OUTLINE: This is a multicenter, cohort study.

Patients are assigned to one of two cohorts according to ECOG performance status (ECOG 0-1 [cohort A] vs ECOG 2 [cohort B]). Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for at least 1 year.

ELIGIBILITY:
Criteria:

* Hemoglobin >= 9 g/dL
* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck:

  * Recurrent and/or metastatic disease
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques OR as >= 10 mm with spiral CT scan
* No known brain metastases
* Life expectancy >= 2 months
* ECOG performance status (PS) 0-1 or Karnofsky PS 70-100% (for patients in cohort A)
* ECOG PS 2 or Karnofsky PS 60-70% (for patients in cohort B)
* WBC >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Calcium =< 12.0 mg/dL
* Bilirubin normal
* AST and ALT =< 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance >= 60 mL/min
* QTc < 500 msec
* No New York Heart Association class III or IV heart failure:

  * Patients with the following are eligible provided they have New York Heart Association class II cardiac function on baseline ECHO/MUGA:

    * History of class II heart failure and asymptomatic on treatment
    * Prior anthracycline exposure
    * Prior central thoracic radiation that included the heart in the radiotherapy port
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions to compounds of similar chemical or biological composition to sunitinib malate
* No history of serious ventricular arrhythmia (i.e., ventricular fibrillation or ventricular tachycardia >= 3 beats in a row)
* No history of other significant ECG abnormalities
* No uncontrolled hypertension (defined as systolic blood pressure [BP] >= 140 mm Hg or diastolic BP >= 90 mm Hg)
* No condition resulting in an inability to take oral medication, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
  * Active peptic ulcer disease
* No gastrostomy, jejunostomy, or other forms of enteral tube-feeding modalities
* No serious or nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No cerebrovascular accident or transient ischemic attack within the past 12 months
* No myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within the past 12 months
* No pulmonary embolism within the past 12 months
* No pre-existing uncontrolled thyroid abnormality (i.e., inability to maintain thyroid function within the normal range with medication)
* No uncontrolled intercurrent illness, including either of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situation that would limit compliance with study requirement
* No more than two prior regimens for recurrent or metastatic disease:

  * Prior chemotherapy as part of initial curative intent therapy (e.g., neoadjuvant, adjuvant, or concurrent chemoradiotherapy) is allowed and will not count as prior therapy for recurrent or metastatic disease
* At least 4 weeks since prior major surgery
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 4 weeks since prior radiotherapy
* No prior treatment with any other antiangiogenic agent (e.g., bevacizumab, sorafenib, pazopanib, AZD2171, vatalanib, or VEGF Trap)
* No prior surgical procedure affecting absorption
* At least 7 days since prior and no concurrent use of CYP3A4 inhibitors, including any of the following:

  * Azole antifungals (e.g., ketoconazole, itraconazole)
  * Verapamil
  * Clarithromycin
  * HIV protease inhibitors (e.g., indinavir, saquinavir, ritonavir, atazanavir, nelfinavir)
  * Erythromycin
  * Delavirdine
  * Diltiazem
* At least 12 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Phenytoin
  * Rifabutin
  * Hypericum perforatum (St. John's wort)
  * Carbamazepine
  * Efavirenz
  * Phenobarbital
  * Tipranavir
* No concurrent therapeutic doses of coumarin-derivative anticoagulants (e.g., warfarin):

Concurrent dosing of =< 2 mg of warfarin daily for prophylaxis of thrombosis is allowed; Concurrent low molecular weight heparin allowed provided prothrombin time INR is =< 1.5

* No other concurrent investigational agents
* No concurrent agents with proarrhythmic potential, including any of the following:

  * Terfenadine
  * Quinidine
  * Procainamide
  * Disopyramide
  * Sotalol
  * Probucol
  * Bepridil
  * Haloperidol
  * Risperidone
  * Indapamide
  * Flecainide
* No other concurrent anticancer agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib -- Cohort A: Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. ECOG Performance Status 0 -1.
- Sunitinib -- Cohort B: Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.ECOG Performance Status 2.
Period: Overall Study
Arm/Group | Sunitinib -- Cohort A | Sunitinib -- Cohort B
Started | 15 | 7
Completed | 15 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib -- Cohort B: Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. ECOG Performance Status 2.
- Total: Total of all reporting groups
Arm/Group | Sunitinib -- Cohort A | Sunitinib -- Cohort B | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Continuous [Median (Full Range); unit: years] | 55 (43-78) [43 to 78] | 60 [40 to 77] | 57 [40 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate (Complete Response [CR] and Partial Response [PR]) Using RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: While patient remains on treatment, up to 30 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Sunitinib -- Cohort A; Sunitinib -- Cohort B: Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Sunitinib -- Cohort A | Sunitinib -- Cohort B
Number analyzed (Participants) | 15 | 7
percentage of participants | 6.7 [0.2 to 31.9] | 0 [0 to 41.0]

2. Primary Outcome: Feasibility of Treatment
Description: Ability to remain on treatment without dose reduction
Time Frame: While patient remains on treatment, up to 30 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib -- Cohort A | Sunitinib -- Cohort B
Number analyzed (Participants) | 15 | 7
percentage of participants | 80.0 [51.9 to 95.7] | 71.4 [29.0 to 96.3]

3. Secondary Outcome: Progression-free Survival
Description: Time to disease progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Sunitinib -- Cohort A | Sunitinib -- Cohort B
Number analyzed (Participants) | 15 | 7
weeks | 8.4 [3 to 26] | 10.5 [3 to 30]

4. Secondary Outcome: Overall Survival
Description: Time from start of treatment until death from any cause.
Time Frame: Up to two years
Measure: Median (Full Range); unit: weeks
Arm/Group | Sunitinib -- Cohort A | Sunitinib -- Cohort B
Number analyzed (Participants) | 15 | 7
weeks | 21.1 [4 to 96] | 19.1 [2 to 70]

ADVERSE EVENTS:
Time Frame: Up to two years
Description: Common Terminology Criteria for Adverse Events (CTCAE v3.0). Reported are grade 1 or higher adverse events.
Arm/Group | Sunitinib -- Cohort A | Sunitinib -- Cohort B
Serious Adverse Events (participants affected / at risk) | 3/15 | 1/7
Other Adverse Events (participants affected / at risk) | 14/15 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib -- Cohort A (N=15) | Sunitinib -- Cohort B (N=7)
Sudden death from sepsis (Infections and infestations) | 1 | 0
Sudden cardiac death (Cardiac disorders) | 0 | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Grade 2
Pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib -- Cohort A (N=15) | Sunitinib -- Cohort B (N=7)
Neutrophil count decreased (Investigations) | 3 | 1
Leukocytes (Blood and lymphatic system disorders) | 6 | 1
Lymphopenia (Blood and lymphatic system disorders) | 6 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 5 | 3
Fatigue (General disorders) | 11 | 3
Anorexia (Metabolism and nutrition disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 5 | 3
Mucositis (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 5 | 3
Hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0
Headache (Nervous system disorders) | 3 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Tumor hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Alkaline phosphatase increased (Investigations) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anal pain (Gastrointestinal disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 1
Confusion (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 4 | 1
Edema limbs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Edema: head and neck (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 1
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INR increased (Blood and lymphatic system disorders) | 1 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Oral hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oral pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neck soft tissue necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 | 0
Sweating (General disorders) | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Taste alteration (General disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Weight loss (Metabolism and nutrition disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less